CLINICAL TRIAL: NCT06645002
Title: Effect of Short and Long-Term Treatment of Stevia Leave Powder on Blood Glucose and Lipid Profile of Diabetic Patients.
Brief Title: Effect of Stevia Leave Powder on Blood Glucose and Lipid Profile of Diabetic Patients
Acronym: Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: Allied Hospital Faisalabad (Other)
Responsible Party: Principal Investigator, Fasiha Ahsan, PhD scholar, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/774/2020
Record Dates: First submitted 2024-09-27; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Diabetes
Keywords: Diabetes; Stevia; Glucose; Lipid profile
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- short term study (Experimental): short term study (7 days) stevia leave powder 1000 mg/day
  Interventions: Dietary Supplement: stevia rebaudiana bertoni
- long term study (Experimental): Long term study (60 days) stevia leave powder 1000 mg/day
  Interventions: Dietary Supplement: stevia rebaudiana bertoni

INTERVENTIONS:
Dietary Supplement: stevia rebaudiana bertoni — effect of short term study (7 days) of stevia leave powder 1000 mg/day in diabetic subjects
Dietary Supplement: stevia rebaudiana bertoni — effect of long term study (60 days) of stevia leave powder 1000 mg/day in diabetic subjects
  Arms: long term study

SUMMARY:
The goal of this clinical trial is to know if stevia leave powder capsule (1000 mg/day) will work to treat diabetes in participants. The main objectives it aims to answer are:

Does stevia decrease the blood glucose level in diabetic subjects that will use stevia powder capsule? Does stevia play its role in blood lipid profile in diabetic subjects that will use stevia powder capsule? The purpose of the study to see the impact of stevia in short (7 days) and long-term treatments (60 days) in diabetic subjects and compare the results

Diabetic subjects will:

Take stevia powder capsule every day for 7 days in short term study Take stevia powder capsule every day for 60 days in long term study

Check the biochemical assessment including blood glucose and lipid profile tests at 0 and 7th days in short term study Check the biochemical assessment including blood glucose and lipid profile tests at 0 and 30 and 60th days in long term study Keep a record of all the tests for comparison

DETAILED DESCRIPTION:
The selected participants will be randomly divided into placebo and treatment groups. The Initial (0-Day) data on anthropometric measurements and blood analysis on glucose, lipid levels and liver function tests (LFTs) will be carried out.

The balance diet plan will be prepared according to Pakistan dietary guidelines and given to all the study participants. Treatment stevia powder capsules will be provided to the participants for 7 days and for 60 days for short and long-term study respectively, for monitoring of compliance. Anthropometric measurements and biochemical assessments like blood glucose levels, lipid profile, insulin resistance and LFTs for short-term study will be measured at baseline, 7th and 60th day while, measurements of blood glucose, lipid profile, insulin resistance and LFTs will be carried out a baseline, 30, and 60 days for long-term study. In this research we will be analysed the effect of stevia powder capsules on diabetic patients for short and long term study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: Individuals with the following conditions will be included as participants;

* Patients of type 2 diabetes mellitus with the age range between 25-35 years from both genders
* Diabetic patients without anti-diabetic drugs and their duration of diabetes no longer than 6 months
* Diabetic patients with HbA1c >6% and blood sugar level >200 mg/dL

Exclusion Criteria:

Individuals with the following conditions were not included as participants;

* Patients with nephropathy, retinopathy, diabetic foot, phenylketonuria, maple syrup urine disease
* Participants with acute and chronic kidney disease, kidney stone,
* Participants with history of acute liver injury (e.g., hepatitis) or severe cirrhosis
* Diabetic patients with obesity, cardiovascular diseases, pregnancy
* Participants taking nutritional supplements and other medicines

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2025-02-22 (Estimated)

PRIMARY OUTCOMES:
To compare the effects of short and long-term treatment of stevia powder capsules on blood glucose levels among diabetic patients | Short term study (7 days) long term study (60 days)
  Teatment group respondents of short term study will be received the stevia powder capsules of 1000mg for 7 days, this group includes the initial screening and assessment of subjects suffering from type-II diabetes. The subjects will also being studied for medical history and anthropometric parameters which include height and weight, BMI and biochemical parameters which include blood glucose levels of fasting, post-prandial, insulin resistance and HbA1c In addition, a dietary study will also be done by food diary method on 3 alternative days. The biochemical parameters of the subjects will be measured at 0, 7th and at 60th day.
  Long-term treatment group participants will receive the treatment with 1000mg stevia powder in capsulated form once per day for 60 days, this group will also undergo the initial screening and assessment of anthropometric and biochemical parameters at 0, 30th and 60th day then will perform comparison analysis at 60th day for both short and long-term studies.

SECONDARY OUTCOMES:
To compare the effects of short and long-term treatment of stevia powder capsules on lipid profile and LFTs among diabetic patients | Short term study (7 days) long term study (60 days)
  Treatment group respondents of short term study will be received the stevia powder capsules of 1000mg for 7 days, After initial assessment, BMI and blood glucose levels record, the lipid profile including, cholesterol, HDL, LDL and LFTs including ALT, AST will also be measured 0, 7th and at 60th day. Same tests will also be performed on long-term study participants and will measure the results at 0, 30 and 60th day of the study, then will perform comparison analysis at 60th day for both short and long-term studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Allied Hospital Faisalabad, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Primary reason for not sharing the IPD is to protect participants privacy

REFERENCES:
- [Background] Ritu M, Nandini J. Nutritional composition of Stevia rebaudiana, a sweet herb, and its hypoglycaemic and hypolipidaemic effect on patients with non-insulin dependent diabetes mellitus. J Sci Food Agric. 2016 Sep;96(12):4231-4. doi: 10.1002/jsfa.7627. Epub 2016 Feb 22. PMID 26781312